CLINICAL TRIAL: NCT05491421
Title: A Phase 1, Randomized, Parallel Assignment, Double Blind, Placebo Controlled, Single and Multiple Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study of ZT002 in Healthy Participants
Brief Title: A Study of ZT002 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QL Biopharmaceutical Australia Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry); Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Organization: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZT002
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (ZT002) (Experimental): Drug: ZT002
  Dose level:
  SAD dose (Cohort 1-4)
  * 0.03 mg/kg, 0.09 mg/kg, 0.18 mg/kg, 0.3 mg/kg;
  MAD dose (Cohort 1-3)
  * Cohort 1: 7.0mg, 10mg, 20mg;
  * Cohort 2: 10 mg, 20mg, 40mg;
  * Cohort 3: To be decided post safety review meetings
  Dose: Subcutaneous Injection
  Interventions: Drug: ZT002
- B (Placebo) (Placebo Comparator): Dose level:
  SAD dose (Cohort 1-4)
  * 0.03 mg/kg, 0.09 mg/kg, 0.18 mg/kg, 0.3 mg/kg;
  MAD dose (Cohort 1-3)
  * Cohort 1: 7.0mg, 10mg, 20mg;
  * Cohort 2: 10 mg, 20mg, 40mg;
  * Cohort 3: To be decided post safety review meetings
  Dose: Subcutaneous Injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ZT002 — Participants will receive a single subcutaneous (SC) ZT002 dose of 0.03, 0.09, 0.18, or 0.3 mg/kg respectively, for SAD Cohorts 1 to 4 under fasted conditions.
  Participants will MAD Cohorts will receive a single subcutaneous (SC) ZT002 in following doses under fasting conditions-
  * Cohort 1: 7.0mg, 10mg, 20mg;
  * Cohort 2: 10 mg, 20mg, 40mg;
  * Cohort 3: To be decided post safety review meetings
  Arms: A (ZT002)
Other: Placebo — Participants will receive same volume as of the study drug of 0.03, 0.09, 0.18, or 0.3 mg/kg respectively, for SAD Cohorts 1 to 4 under the fasted condition.
  Participants in MAD cohorts will receive same volume as study drug in the following cohorts under fasted condition-
  * Cohort 1: 7.0mg, 10mg, 20mg;
  * Cohort 2: 10 mg, 20mg, 40mg;
  * Cohort 3: To be decided post safety review meetings
  Arms: B (Placebo)

SUMMARY:
This study will comprise a randomized, parallel assignment, double blind, placebo controlled, single and multiple ascending dose, safety, tolerability and pharmacokinetic study of ZT002 in healthy participants.

DETAILED DESCRIPTION:
This study is planned to be conducted in 2 portions: single ascending dose and multiple ascending doses.

For the SAD portion, there are a total of 4 cohorts. In each cohort 6 participants will receive ZT002, and 2 participants will receive placebo, for a total of 8 participants in each cohort.

For the MAD portion, the study is planned to be conducted in healthy participants with a BMI range of 26kg/m^2 to 40kg/m^2 and a body weight of >/= 80kg. This portion is planned to be conducted in 3 cohorts (Cohort 1 to 3), 6 participants will receive ZT002, and 2 participants will receive placebo, across of total of 8 participants (for a total of 24 participants across 3 cohorts). In each cohort, 3 escalating doses of ZT002 are planned. Dosing is planned to be administered every 2 weeks (Q2W).

Potential participants will be screened to assess their eligibility to enter the study in a Screening period from days -28 to -2, prior to the scheduled treatment on Day 1.

A Safety Monitoring Committee (SMC) meeting to discuss dose escalation will be held after each cohort

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-55 years, both inclusive, at time of informed consent
2. Body Mass Index (BMI) between 22.0～35.0 kg/m2 both included. For the MAD portion only, participants with BMI range of 26 kg/m2 to 40 kg/m2 and a body weight of ≥ 80 kg will be included.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations at screening and before administration of study drug, as assessed by the Investigator
4. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.
5. Has no relevant dietary restrictions (not including those common restrictions that can be easily accommodated, i.e., veganism, vegetarianism, halal, etc.), and willing to consume standard meals within the options provided by the site
6. Male participants must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a woman of childbearing potential (WOCBP), the participant must be surgically sterile (>30 days since vasectomy with no viable sperm) or the participant and his partner must be using an acceptable, highly effective contraceptive method from 4 weeks prior to dosing until study completion, including the follow-up period.

   Female participants that are WOCBP must be non-pregnant and non-lactating, and using an acceptable, highly effective contraceptive method from 4 weeks prior to dosing until study completion, including the follow-up period, OR must be abstinent from heterosexual intercourse OR their partner must be surgically sterile (>30 days since vasectomy with no viable sperm), provided the male partner is a sole partner.

   Female participants that are not WOCBP must have documented evidence of surgical sterilization at least 6 months prior to Screening (e.g., hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), OR must be postmenopausal for ≥12 months. Postmenopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female participants.

   Acceptable methods of contraception include the use of condoms AND the use of an effective contraceptive for the female partner that includes: oral contraceptive pill (OCPs), long acting implantable hormones, injectable hormones, contraceptive patches, a vaginal ring or an intrauterine device (IUD).

   Participants with same-sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle, and no contraception is required.
7. Male participants agree not to donate sperm for at least 90 days after the last dose of study drug.

Exclusion Criteria:

1. History of significant drug allergy or drug hypersensitivity.
2. Known or suspected allergy to trial product or related products.
3. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee), that could adversely affect the safety of the participant or their likelihood to comply with the protocol or complete the study per protocol. Fully resolved childhood asthma is not exclusionary. Gestational diabetes is exclusionary.
4. eGFR value ≤90 mL/min/1.73m2 using the MDRD equation.
5. Clinically significant abnormal laboratory test results during the Screening and before administration of study drug, as judged by the Investigator.
6. Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or medullary thyroid carcinoma (MTC) as declared by the participant.
7. History of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
8. History of acute or chronic pancreatitis.
9. Calcitonin equal or above 50 ng/L at screening.
10. Fever (body temperature >37.5°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening and Day -1.
11. History of severe allergic or anaphylactic reactions.
12. QTcF > 450 ms for male participants or > 470 ms for female participants, or any other abnormal ECG findings that are considered by the Investigator to be clinically significant, at Screening and before administration of study drug.
13. History or presence of a condition associated with significant immunosuppression.
14. History of life -threatening infection (e.g. meningitis).
15. Infections requiring parenteral antibiotics within the 6 months prior to Screening.
16. History of drug/chemical substance abuse within 1 year from Screening.
17. Positive alcohol breath test result, or positive urine drug screen (confirmed by repeat), at Screening or check-in.
18. Regular alcohol consumption (by self-declaration) in the past 6 months, defined as greater than 21 alcohol units per week for males and 14 units per week for females (where 1 unit = 284 mL of beer, 25 mL of 40% spirit or a 125 mL glass of wine).

    Unwilling to abstain from alcohol consumption from 24 hours prior to admission to the CRU, during the residency period, and 24 hours prior to each non-residential visit.
19. Have smoked >5 cigarettes or use the equivalent tobacco or nicotine containing products per day in the past 1 month prior to Screening (vaping with nicotine containing vapes included) or unable or unwilling to refrain from smoking and use of nicotine substitute products until after the final study visit, as judged by the Investigator.
20. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening.
21. Previously dosed in a clinical trial involving this or other IPs within the last 3 months before dosing.
22. Blood donation or considerable blood loss - more than 400 mL, during the 3 months prior to study start, and plasma donation within 7 days prior to study start.
23. Systolic blood pressure >140 or <90 mmHg, diastolic blood pressure >90 or <40 mmHg, and pulse rate >100 or <40 beats per minute. Abnormal values should be confirmed by a repeat measurement (one repeat only).
24. Impaired hepatic function measured as ALT (Alanine aminotransferase), AST (Aspartate aminotransferase), alkaline phosphatase above 1.5 times the upper reference limit (one retest of the initial test is permitted, the last result being conclusive).
25. Confirmed diagnosis of diabetes mellitus type 1, type 2, or of any other forms at any time, and/or occurrence of documented or suspected hypoglycemic episodes within 12 months prior to Screening, and any current or prior use of insulin secretagogues (e.g., sulfonylurea) or insulin.
26. Impaired glucose tolerance results for oral glucose tolerance test (OGTT) performed at screening. A blood glucose level ≥7.8 mmol/L at 2 hours will be considered as impaired glucose tolerance.
27. Those who have been vaccinated within 4 weeks prior to screening or who are scheduled to be vaccinated within 4 weeks of dosing, except for COVID-19 and influenza vaccines, exclusionary when the participant is scheduled to be vaccinated within 1 week of dosing.
28. Exposure to any significantly immune suppressing drug (including experimental therapies as part of a clinical trial) within the 4 months prior to Screening or 5 half-lives, whichever is longer.
29. Use of prescription or non-prescription systemic or topical medicinal products (except routine vitamins, supplements, acetylsalicylic acid, paracetamol and contraceptives; herbal preparations or dietary supplements that are specifically marketed for control of body weight or appetite remain excluded) within 3 weeks (or within 5 half-lives of the medicinal product, whichever is longest) prior to the dosing and for the duration of the study. Paracetamol/acetaminophen (1-2 therapeutic doses per week) may be used for minor ailments during the course of the study, at the discretion of the Investigator.
30. Poor peripheral venous access.
31. Participant is unwilling to refrain from strenuous exercise (including weightlifting) from 48 hours prior to admission to the investigational site until completion of the residency (inpatient) period, and from 48 hours prior to the Day 15, Day 29, Day 43, and Day 71/Early Withdrawal visits.
32. Any disorder or other circumstance which in the Investigator's opinion might jeopardize participant's safety, evaluation of results, or compliance with the protocol, meaning that, in the opinion of the Investigator (or designee), the participant should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single escalation dose of ZT002 through the incidence and severity of treatment emergent adverse events in SAD Cohorts. Number of participants with treatment-emergent adverse events. | Up to 71 days
  Coded by the most updated version of the Medical Dictionary for Regulatory Activities (MedDRA).
Safety and tolerability of a single escalation dose of ZT002 through the incidence severity of serious adverse events in SAD Cohorts. Number of participants with serious adverse events. | Up to 71 days
  Coded by the most updated version of the Medical Dictionary for Regulatory Activities (MedDRA).
To assess safety and tolerability of multiple escalation doses of ZT002 in healthy participants with a BMI range of 26 kg/m2 to 40 kg/m2 and a body weight of ≥80 kg through number of participants with treatment emergent adverse events in MAD Cohorts. | up to 85 days
  Coded by the most updated version of the Medical Dictionary for Regulatory Activities (MedDRA).
To assess safety and tolerability of multiple escalation doses of ZT002 in healthy participants with a BMI range of 26 kg/m2 to 40 kg/m2 and a body weight of ≥80 kg through incidence severity of serious adverse events in MAD Cohorts. | Upto 85 days
  Coded by the most updated version of the Medical Dictionary for Regulatory Activities (MedDRA).

SECONDARY OUTCOMES:
The Pharmacokinetics (PK) profile of a single escalation dose of ZT002 in healthy participants in SAD and MAD Cohorts. Parameter: Maximum observed plasma concentration of ZT002 (Cmax) | Up to 85 days
The Pharmacokinetics (PK) profile of a single escalation dose of ZT002 in healthy participants in SAD and MAD Cohorts. Parameter: Area under the drug-time curve from 0 h after dosing to the last quantifiable concentration time point (AUC0-last) | Up to 85 days
The Pharmacokinetics (PK) profile of a single escalation dose of ZT002 in healthy participants in SAD and MAD cohorts. Parameter: Area under the drug-time curve to infinity (AUC0-inf) | Up to 85 days
The anti-drug antibody (ADA) response through an anti-drug antibody assay in SAD and MAD cohorts. | Up to 85 days
The anti-drug antibody (ADA) response through testing serum or plasma of the participant post dosing in SAD and MAD cohorts. | Up to 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Q-Pharm Pty Limited, Herston, Queensland, Australia